CLINICAL TRIAL: NCT02178852
Title: Effect of Trigeminal Nerve Stimulation (TNS) on Nicotine Craving: Phase II, Cross-over, Randomized, Sham-controlled Clinical Trial
Brief Title: TNS for Treating Nicotine Craving
Acronym: TNS-nicotine
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Santa Casa Medical School (Other)
Responsible Party: Principal Investigator, Pedro Shiozawa, Coordinator Neuromodulation Laboratory, Santa Casa Medical School
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNS-nicotine
Record Dates: First submitted 2014-06-26; First posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Nicotine Craving

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TNS-active (Experimental): TRIGEMINAL NERVE STIMULATION (TNS)
  Interventions: Device: TRIGEMINAL NERVE STIMULATION (TNS)
- TNS-sham (Placebo Comparator): TRIGEMINAL NERVE STIMULATION (TNS) - sham

INTERVENTIONS:
Device: TRIGEMINAL NERVE STIMULATION (TNS) — TNS stimulation over V1 branches of V cranial nerve. Single session for 30 minutes. The patient will undergo a specific cue-induced cigarette craving model during the final 3 minutes of stimulation. Craving scores will be rated before and after stimulation
  Other Names: TNS
  Arms: TNS-active

SUMMARY:
Electrical stimulation provides direct modulatory effects on subcortical regions. Indeed, neuroimaging studies show changes in neural activity in specific brain regions such as the amygdala, insula, precentral gyrus, hippocampus and thalamus. The neuroanatomical connections established with the trigeminal nerve have been associated with the mechanism called "bottom-up" neuromodulation. According to this hypothesis, the spread of electrical stimulation follows a path from the peripheral nerves towards the brain stem was then advertise for cortical and subcortical regions. Connections to structures involved in the reward system as the amygdala and hippocampus could theoretically modulate dysfunctional brain activity in these regions, which may induce favorable clinical effects.

ELIGIBILITY:
Inclusion Criteria:

1. patients over 18 years
2. both genres
3. diagnosed with nicotine related disorder for at least 12 months according to the diagnostic criteria of DSM-IV administered by a psychiatrist.
4. Also we will adopt as inclusion criteria a score of Nicotine Dependence Fagerstrom Test greater or equal to 5 points.
5. Finally, patients should be able to read and understand the portuguese language.
6. Patients will be selected from spontaneous demand. In accordance to informed consent -

Exclusion Criteria:

1. other psychiatric diagnosis such as bipolar Affective Disorder, alcohol dependence, schizophrenia and dementia.
2. Also excluded patients with severe neurological or medical diseases, such as neurodegenerative diseases, stroke, cancer in activity, congestive heart failure or chronic obstructive pulmonary disease stage III or IV.
3. Finally, patients with severe suicidal ideation (structured planning suicide or attempted suicide in the past 4 weeks) will be excluded. In this case, the patient will be seen immediately by a psychiatrist of the research itself that will take the appropriate clinical management according to the severity of suicidal thinking.

   -

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Craving for nicotine | (T1) Immediately before TNS protocol ; (T2) 30 minutes after TNS protocol
  Craving for nicotine assessed by visual scale before and after cue-induced images for nicotine craving. Patients will be exposed to visual model for cue-induced images related to nicotine craving during the last 3 minutes of the TNS protocol (which has an overall time of 30 minutes). Main comparison will be between T1 and T2 craving level.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Shiozawa, MD, Principal Investigator — Neuromodulation Laboratory - Santa Casa Medical School; Pedro Shiozawa, MD, Study Director — Neuromodulation Laboratory - Santa Casa Medical School; Quirino Cordeiro, MD PhD, Study Chair — Neuromodulation Laboratory - Santa Casa Medical School
Locations (1):
- Centro de Atencao Integrada à Saúde Mental - CAISM, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Fecteau S, Agosta S, Hone-Blanchet A, Fregni F, Boggio P, Ciraulo D, Pascual-Leone A. Modulation of smoking and decision-making behaviors with transcranial direct current stimulation in tobacco smokers: a preliminary study. Drug Alcohol Depend. 2014 Jul 1;140:78-84. doi: 10.1016/j.drugalcdep.2014.03.036. Epub 2014 Apr 16. PMID 24814566
- [Background] Luigjes J, Breteler R, Vanneste S, de Ridder D. [Neuromodulation as an intervention for addiction: overview and future prospects]. Tijdschr Psychiatr. 2013;55(11):841-52. Dutch. PMID 24242143
- [Background] Pedron S, Monnin J, Haffen E, Sechter D, Van Waes V. Repeated transcranial direct current stimulation prevents abnormal behaviors associated with abstinence from chronic nicotine consumption. Neuropsychopharmacology. 2014 Mar;39(4):981-8. doi: 10.1038/npp.2013.298. Epub 2013 Oct 24. PMID 24154668
- [Background] Xu J, Fregni F, Brody AL, Rahman AS. Transcranial direct current stimulation reduces negative affect but not cigarette craving in overnight abstinent smokers. Front Psychiatry. 2013 Sep 20;4:112. doi: 10.3389/fpsyt.2013.00112. eCollection 2013. PMID 24065930
- [Background] Grundey J, Thirugnanasambandam N, Kaminsky K, Drees A, Skwirba AC, Lang N, Paulus W, Nitsche MA. Rapid effect of nicotine intake on neuroplasticity in non-smoking humans. Front Pharmacol. 2012 Oct 26;3:186. doi: 10.3389/fphar.2012.00186. eCollection 2012. PMID 23133419